CLINICAL TRIAL: NCT04405258
Title: Randomized Clinical Trial of Additional Left Atrial Posterior Wall Isolation for Persistent Atrial Fibrillation
Brief Title: Left Atrial Posterior Wall Additional Isolation for Persistent Atrial Fibrillation Trial
Acronym: LEAP-AF
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Institute for Clinical Effectiveness, Japan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 947
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Persistent Atrial Fibrillation; Catheter Ablation; Pulmonary Vein Isolation; Posterior Wall Isolation
Keywords: Persistent atrial fibrillation; Catheter ablation; Pulmonary vein isolation; Posterior wall isolation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVI alone (Active Comparator): Pulmonary vein isolation, superior vena cava isolation, and cavotricuspid isthmus ablation
  Interventions: Procedure: Pulmonary vein isolation
- PVI and PWI (Active Comparator): Pulmonary vein isolation, superior vena cava isolation, cavotricuspid isthmus ablation, and left posterior wall isolation
  Interventions: Procedure: Left posterior wall isolation

INTERVENTIONS:
Procedure: Pulmonary vein isolation — Pulmonary vein isolation, superior vena cava isolation, and cavotricuspid isthmus ablation
  Arms: PVI alone
Procedure: Left posterior wall isolation — Pulmonary vein isolation, superior vena cava isolation, cavotricuspid isthmus ablation, and left posterior wall isolation
  Arms: PVI and PWI

SUMMARY:
The purpose for this study is to determine whether left posterior wall isolation (PWI) in addition to pulmonary vein isolation (PVI) is effective as ablation strategy for persistent atrial fibrillation (AF).

DETAILED DESCRIPTION:
PVI is cornerstone of AF ablation. However, clinical outcome of only PVI in patients with persistent AF is insufficient due to AF substrate extending to left atrium. Strategy of catheter ablation for persistent AF is not established despite attempts of numerous left atrial substrate modifications. Additional PWI on PVI is one of expected effective strategies for persistent AF, because PW originated from common tissue of PV and is considered to play a part in AF trigger and maintenance. However, this strategy is also not established in the recent international consensus statement. Following two reasons are considered. One is the procedural difficulty in creating durable PWI, and another is the existence of patients who can recover by only PVI. The latest technology, ablation index, can create durable PVI, and may create durable PWI. Several reports suggested that PVI only strategy was sufficient in the patients with persistent AF who could maintain sinus rhythm after pharmacological or electrical cardioversion. Therefore, we planed this randomized clinical trial that compared between PVI alone and additional PWI on PVI using ablation index in the patients with persistent AF without pharmacological sinus rhythm conversion.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for first catheter ablation of persistent atrial fibrillation
* Patients without conversion to sinus rhythm within 30 days after antiarrhythmic drug administration
* Patients with persisting duration of atrial fibrillation less than 3 years
* Patients with left atrial diameter less than 50mm
* Patients who can be followed up for 18 months
* Patients with written informed consent

Exclusion Criteria:

* Patients who can not be received adequate anticoagulation therapy
* Patients with history of myocardial infarction within 6 months
* Patients with history of open heart surgery
* Patients scheduled for open heart surgery
* Patients with severe valvular heart disease
* Patients during pregnancy
* Patients with expected life expectancy less than 1 year due to malignancy or non-cardiovascular disease
* Patients considered unsuitable for study by the attending physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial tachyarrhythmia after 90-day blanking period of catheter ablation | 18 months
  Recurrence of atrial tachyarrhythmia is defined atrial arrhythmia that needs admission, electrical cardioversion, and antiarrhythmic drug administration, and/or that persists more than 30 seconds.

SECONDARY OUTCOMES:
Recurrence of atrial fibrillation or atrial tachycardia after 90-day blanking period of catheter ablation | 18 months
  Recurrence of atrial fibrillation or atrial tachycardia needs admission, electrical cardioversion, and antiarrhythmic drug administration, and/or that persists more than 30 seconds.
Recurrence of atrial fibrillation or atrial tachycardia within 90-day after catheter ablation | 90 days
  Recurrence of atrial fibrillation or atrial tachycardia needs admission, electrical cardioversion, and antiarrhythmic drug administration, and/or that persists more than 30 seconds.
Repeated ablation of atrial tachyarrhythmia | 18 months
Recurrence of atrial fibrillation or atrial tachycardia after 90-day blanking period of repeated ablation | 18 months
Atrial Fibrillation Quality of Life Questionnaire | 18 months
  Atrial Fibrillation Quality of Life Questionnaire
Complications of ablation procedure | 1 month
  Complications of ablation procedure includes death, cardiac tamponade, pericardial effusion, systemic embolism, symptomatic strokes, hematoma, A-V shunt, pericarditis, phrenic nerve paralysis, A-V block, procedure-related infections, heart failure, atrio-esophageal fistula, esophageal vagus nerve injury

CONTACTS AND LOCATIONS:
Overall Officials: Keisuke Okawa, MD, Principal Investigator — Kagawa Prefectural Central Hospital
Locations (1):
- Kagawa Prefectural Central Hospital, Takamatsu, Kagawa-ken, Japan

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study will be available from the data center upon reasonable request.